CLINICAL TRIAL: NCT03798483
Title: Individualised Exercise for Adults With an Acute Lateral Patellar Dislocation: a Feasibility Study
Brief Title: INDividualised EXercise for Kneecap Dislocations
Acronym: INDEX-KD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRes/18-19/04/2; 251913 (Other: Health Research Authority - IRAS ID)
Record Dates: First submitted 2018-12-11; First posted 2019-01-10 (Actual); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2018-12

CONDITIONS: Patella Dislocation; Patella Dislocation Recurrent
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized exercise (Experimental): Participants after a lateral kneecap dislocation will be enrolled into an individualized exercise intervention supervised by a physiotherapist
  Interventions: Other: Individualised exercise

INTERVENTIONS:
Other: Individualised exercise — The intervention will be comprised of up to 6, one-to-one physiotherapy sessions, over a maximum duration of 3 months. 1 or 2 extra sessions are allowed if deemed essential by the participant's physiotherapist. Less than 6 physiotherapy sessions can be agreed with the participant if they have achieved their goals. Throughout this time participants will be required to perform an exercise programme a minimum of 3 times per week. The exercise programme aims to increase leg muscle strength and facilitate a return to the participant's usual activities. It may include hopping and change of direction tasks if these are activities the participant would normally do. Behavioural change techniques to increase participant adherence to the exercise programme will also be used.

SUMMARY:
This study is a feasibility study. It will assess areas of uncertainty relating to the implementation of an individualised exercise programme for patients with a recent kneecap dislocation. This will help determine if a future larger study is feasible, and inform the design and conduct of future research that would aim to optimise outcomes after a kneecap dislocation.

DETAILED DESCRIPTION:
The investigators aim to recruit 15 adult participants with a recent, first-time or recurrent kneecap dislocation, from an acute hospital. Participants will receive up to 6 physiotherapy sessions over 3 months. The investigator's exercise programme aims to improve leg muscle strength and facilitate a return to the participant's usual activities. This may include activities such as hopping and changing direction which differentiates it from other programmes. Participants will be required to perform the exercise programme 3 times a week independently. Strategies to increase adherence to the exercise programme will also be used. This study is part of a Masters in Clinical Research funded by the National Institute for Health Research

ELIGIBILITY:
Inclusion Criteria:

* First time or recurrent lateral patella dislocation meeting the diagnostic criteria of 1) requiring reduction by paramedics or 2) diagnosed by a member of the trauma and orthopaedic team.

Exclusion Criteria:

* Concurrent anterior cruciate ligament or posterior cruciate ligament injury confirmed by negative Lachman's and posterior drawer test or confirmed by Magnetic Resonance Imagery (MRI); medial collateral and lateral collateral ligament injury requiring application of a hinged knee brace or surgical repair; concomitant injury that would prohibit participation in the exercise intervention
* > 4 weeks from injury to presentation to acute care (ED or trauma services)
* Unable to give written informed consent
* Previous surgery on the affected knee
* Presence of fracture on plain radiograph including osteochondral fractures
* Medial patellar dislocation
* Considered inappropriate for referral to physiotherapy (by member of trauma and orthopaedic team assessing the patient)
* History of severe neuromuscular or congenital disorders
* Patients referred for orthopaedic opinion who are subsequently listed for surgery prior to completion of the study intervention
* Unable to understand written or spoken English
* Unable to attend physiotherapy sessions at the John Radcliffe trauma outpatient physiotherapy department

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Haddad, PhD, Principal Investigator — City, University of London
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Forde C, Haddad M, Hirani SP, Keene DJ. Is an individually tailored programme of intense leg resistance and dynamic exercise acceptable to adults with an acute lateral patellar dislocation? A feasibility study. Pilot Feasibility Stud. 2021 Nov 8;7(1):197. doi: 10.1186/s40814-021-00932-x. PMID 34749823

RESULTS

PARTICIPANT FLOW:
Groups:
- Individualized Exercise: Participants after a lateral kneecap dislocation were enrolled into an individualized exercise intervention supervised by a physiotherapist
  Participants received up to six, one-to-one, face-to-face physiotherapy sessions, over a maximum duration of 3 months. Less than six physiotherapy sessions were used if participants achieved their goals, were self-managing effectively, and their physiotherapist agreed. Participants had to perform prescribed exercises a minimum of 3 times per week. Prescribed exercise aimed to restore leg muscle strength through intense leg strengthening exercises, and restore activity levels by prescribing dynamic exercises related to the activities participants wished to resume. Behavioural change techniques to increase participant adherence to the exercise programme were also used.
Period: Overall Study
Arm/Group | Individualized Exercise
Started | 15
Returned All Follow-up Outcome Data | 11
Completed (Completed participants were participants that returned Lysholm Knee Scoring Scale data. 2 participants returned Lysholm Knee Scoring Scale outcome data only.) | 13
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Individualized Exercise
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 22 [19 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White British | 13
  Ethnicity: White Other | 1
  Ethnicity: Other | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15
Height [Median (Inter-Quartile Range); unit: meters] | 1.75 [1.62 to 1.8]
Weight [Median (Inter-Quartile Range); unit: Kilograms] | 69.9 [64 to 85]
Education [Count of Participants; unit: Participants]
  Secondary education | 9
  Higher professional or University education | 6
Employment status [Count of Participants; unit: Participants]
  Employed | 12
  Student | 3
Duration from injury to eligibility assessment [Mean (Inter-Quartile Range); unit: days] | 2 [1 to 9]
Previous ipsilateral patellar dislocation [Count of Participants; unit: Participants] | 5
Number of previous ipsilateral patellar dislocations [Count of Participants; unit: Participants]
  0 | 10
  1 | 1
  2 | 1
  3 | 1
  4 | 1
  5-6 | 1
Previous contralateral patellar dislocation [Count of Participants; unit: Participants] | 3
Number of previous contralateral patellar dislocations (number of participants) [Count of Participants; unit: Participants]
  0 | 12
  1 | 1
  2 | 1
  >10 | 1
Family history of patellar dislocation [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Eligibility Rate
Description: Percentage of patients with a diagnosed lateral patellar dislocation, screened for eligibility, who satisfied the eligibility criteria
Time Frame: 15 weeks
Population: These were patients with a clinically diagnosed lateral patellar dislocation who underwent an eligibility assessment
Measure: Count of Participants; unit: Participants
Groups:
- Patients With a Diagnosed Lateral Patellar Dislocation: Patients with a clinically diagnosed lateral patellar dislocation
Arm/Group | Patients With a Diagnosed Lateral Patellar Dislocation
Number analyzed (Participants) | 22
Participants | 15

2. Primary Outcome: Recruitment Rate
Description: Percentage of eligible participants who consented to participate in the study
Time Frame: 15 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Exercise
Number analyzed (Participants) | 15
Participants | 15

3. Primary Outcome: Attrition
Description: Percentage (0-100%) of participants enrolled in the study who failed to provide any 12 week follow-up data
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Exercise
Number analyzed (Participants) | 15
Participants | 2

4. Primary Outcome: Acceptability [Participant Satisfaction]: Questionnaire
Description: Participant response to an internally designed patient questionnaire. This will measure several domains of of intervention acceptability: satisfaction with treatment, self-efficacy, burden of treatment, and intention to adhere. 6 questions will assess satisfaction with treatment, 3 questions will assess self-efficacy,1 question will assess burden of treatment and 1 question will assess intention to adhere. Each question will use a 5 point likert scale (0-4) with lower scores indicating higher satisfaction, self-efficacy, and intention to adhere. Each question will be reported individually.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Participants Who Completed and Returned Follow-up Outcome Data: 11/15 participants completed and returned all follow-up data. The results represents outcome data from these eleven participants
Arm/Group | Participants Who Completed and Returned Follow-up Outcome Data
Number analyzed (Participants) | 11
units on a scale
  How satisfied are you with the effect of your physiotherapy treatment? | 0 [0 to 0]
  How satisfied are you with your involvement in decision making about your physiotherapy treatment? | 0 [0 to 0]
  How satisfied were you with up to six physiotherapy sessions over three months after your injury? | 0 [0 to 0]
  How satisfied were you with the written information you were given describing the study? | 0 [0 to 0]
  How satisfied were you with the written information you were given about your injury? | 0 [0 to 1]
  How satisfied are you overall with the physiotherapy care you received after your injury? | 0 [0 to 0]
  How confident are you that you can return to all your normal activities? | 0 [0 to 1]
  How did doing your exercises fit into your weekly routine? | 1 [0 to 2]
  How confident are you that you were doing your exercises the way your physiotherapist showed you? | 1 [0 to 1]
  How confident are you that you understood how tiring the muscle strengthening exercises should feel? | 1 [0 to 1]
  How likely are you to continue your exercises now your physiotherapy is finished? | 1 [0 to 1]

5. Primary Outcome: Adherence
Description: Percentage (0-100%) of scheduled physiotherapy sessions attended
Time Frame: 12 weeks
Measure: Count of Units; unit: Scheduled physiotherapy sessions
Units Other Than Participants: Scheduled physiotherapy sessions
Arm/Group | Individualized Exercise
Number analyzed (Participants) | 15
Number analyzed (Scheduled physiotherapy sessions) | 66
Scheduled physiotherapy sessions | 56

6. Primary Outcome: Adherence [Participant-reported Adherence to Home Exercise Using a Likert Scale]
Description: Participant response at follow-up to the question 'how often did you perform your exercises at least three times a week?' using a five-point Likert scale (0-4) anchored at 'always' (0) and 'never' (4)
Time Frame: 12 weeks
Population: 11/15 participants completed and returned data for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Completed and Returned Follow-up Outcome Data
Number analyzed (Participants) | 11
Participants
  'Always' | 4
  'Often' | 5
  'Sometimes' | 2

7. Secondary Outcome: Acceptability of Outcome Data Collection
Description: Percentage (0-100%) of questions completed in the following patient-reported outcome measures: Lysholm Knee Scoring Scale, Tegner Activity Scale, EQ-5D-5L, completed at baseline and returned at 3-month follow-up
Time Frame: 12 weeks
Population: 15 participants completed baseline patient-reported outcome measures and 11 participants completed all patient-reported outcome measures at 3-month follow-up and returned by post. Analysed data refers only to these participants.
  Lysholm Knee Scoring Scale outcome data was obtained for 2 participants by phone at 3-month follow-up, so they are not included in analysed data
Measure: Number; unit: percentage of questions
Arm/Group | Individualized Exercise
Number analyzed (Participants) | 15
percentage of questions
  Baseline Lysholm Knee Scoring Scale | 100
  Baseline Tegner Activity Scale | 100
  Baseline EQ-5D-5L | 100
  Follow-up Lysholm Knee Scoring Scale: number analyzed (Participants) | 11
  Follow-up Lysholm Knee Scoring Scale | 100
  Follow-up Tegner Activity Scale: number analyzed (Participants) | 11
  Follow-up Tegner Activity Scale | 100
  Follow-up EQ-5D-5L: number analyzed (Participants) | 11
  Follow-up EQ-5D-5L | 100

8. Secondary Outcome: Number of Treatment Related Adverse Events Experienced by Participants
Description: The total number and type of treatment related adverse events experienced by participants will be recorded. This will be recorded from commencement of the intervention to 12 week follow-up. Treatment related adverse events will be recorded by physiotherapists at each physiotherapy session and by participant self report at 12 week follow up.
Time Frame: Through 12 weeks after first physiotherapy session
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Exercise
Number analyzed (Participants) | 15
Participants
  knee pain or swelling after completing prescribed exercises that lasted >1 week | 1
  Recurrent patella dislocation | 1
  No treatment related adverse event | 13

9. Secondary Outcome: Presence/Absence of Common Lateral Patella Dislocation Diagnostic Criteria
Description: Following diagnosis of a lateral patellar dislocation by an orthopaedic surgeon or physiotherapist, the clinician will be asked which of the following proposed assessment findings to include in the eligibility criteria for future studies, were present/absent during their clinical examination: positive patella apprehension test, visible knee joint effusion or haemarthrosis, medial patellofemoral ligament tenderness on palpation, and a convincing patient history of a visible deformity on the lateral aspect of the knee or a sensation of the patella 'popping' out of joint followed by spontaneous reduction
Time Frame: Baseline
Population: 15 participants were assessed for all the clinical findings below, except for the patella apprehension test which was only assessed in 13 participants.
Measure: Number; unit: percentage
Arm/Group | Patients With a Diagnosed Lateral Patellar Dislocation
Number analyzed (Participants) | 15
percentage
  Medial patellofemoral ligament tenderness | 100
  convincing history of a lateral patellar dislocation | 93.3
  visible knee joint effusion or haemarthrosis | 66.7
  positive patella apprehension test,: number analyzed (Participants) | 13
  positive patella apprehension test, | 100

10. Secondary Outcome: Tegner Activity Scale Questionnaire
Description: This measures activity on a scale from 0-10, with higher scores indicating higher activity. It will be administered as a patient completed questionnaire.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Participants Who Completed and Returned Follow-up Outcome Data
Number analyzed (Participants) | 11
units on a scale | 6 [3 to 7]

11. Secondary Outcome: Lyhsolm Knee Scoring Scale Questionnaire
Description: It is scored from 0-100 with lower scores indicating higher pain and disability. It will be administered as a patient completed questionnaire.
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Patients Who Returned Lysholm Knee Scoring Scale Outcome Data: 13 participants returned Lysholm Knee Scoring Scale data, for 2 of these participants outcome data was obtained by phone
Arm/Group | Patients Who Returned Lysholm Knee Scoring Scale Outcome Data
Number analyzed (Participants) | 13
units on a scale | 90 [76.5 to 95]

12. Secondary Outcome: Quality of Life Using the EQ-5D-5L Questionnaire
Description: This assess quality of life using 5 domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depress, each containing 5 options. These domains are combined to give a single score ranging from -0.594 to 1 for UK populations, with higher scores indicating higher quality of life. Participants rate their overall health on a visual analogue scale from 0 (worst health you can imagine) to 100 (the best help you can imagine). It will be administered as a patient completed questionnaire.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Participants Who Completed and Returned Follow-up Outcome Data
Number analyzed (Participants) | 11
units on a scale
  Index score | 0.84 [0.8 to 1]
  Health on a Visual Analogue Scale | 90 [85 to 95]

13. Secondary Outcome: Assess Delivery of the Intervention [Duration From Injury to Commencing Physiotherapy]
Description: Treatment logs will be analysed to record the duration (number of days) from injury to commencing the intervention
Time Frame: From date of injury until date of the first physiotherapy session, assessed up to 6 weeks
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Individualized Exercise
Number analyzed (Participants) | 15
Days | 21 [15 to 27]

14. Secondary Outcome: Assess Delivery of the Intervention [Number of Physiotherapy Sessions Received by Participants]
Description: Treatment logs will be analysed to assess the number of physiotherapy sessions received by participants
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: physiotherapy sessions
Arm/Group | Individualized Exercise
Number analyzed (Participants) | 15
physiotherapy sessions | 3 [3 to 5]

15. Secondary Outcome: Assess Delivery of the Intervention [Duration of Intervention]
Description: Treatment logs will be analysed to assess the duration (days) of the study intervention
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Individualized Exercise
Number analyzed (Participants) | 15
Days | 50 [37 to 79]

16. Secondary Outcome: Assess Delivery of the Intervention [Types of Exercises Prescribed by Physiotherapists]
Description: Treatment logs will be analysed to assess the types of exercise prescribed by physiotherapists to participants
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Individualized Exercise
Number analyzed (Participants) | 15
participants
  Knee flexibility exercise | 13
  Trunk and leg control exercise | 14
  Leg resistance exercise | 15
  Running exercise | 5
  Bespoke exercise | 5

17. Secondary Outcome: Assess Delivery of the Intervention [Dose of Exercises Prescribed by Physiotherapists]
Description: Treatment logs will be analysed to assess the dose of exercise prescribed by physiotherapists to participants
Time Frame: 12 weeks
Measure: Count of Units; unit: Prescribed leg resistance exercise
Units Other Than Participants: Prescribed leg resistance exercise
Arm/Group | Individualized Exercise
Number analyzed (Participants) | 15
Number analyzed (Prescribed leg resistance exercise) | 93
Prescribed leg resistance exercise
  Prescribed sets between 1-3 | 90
  Prescribed repetitions between 8-12 | 89
  Prescribed frequency 3 or more per week | 91

18. Secondary Outcome: Assess Delivery of the Intervention [Initial Injury Management]
Description: Treatment logs will be analysed to assess how participants are initially managed by trauma and orthopaedic team
Time Frame: From date of review by trauma and orthopaedic team until date of the first physiotherapy session, assessed up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Exercise
Number analyzed (Participants) | 15
Participants
  Lateral butress splint | 12
  Cricket pad splint | 2
  Hinged knee brace | 1
  Full weight-bearing | 15
  Two elbow crutches | 7
  No walking aids | 8
  Knee range of movement exercises | 7
  Non-weight bearing knee strengthening exercise | 4
  Gait practice, balance exercises | 2
  Weight-bearing knee strengthening, strengthening of unijured joints | 1

ADVERSE EVENTS:
Time Frame: through 3 months after the first physiotherapy session
Arm/Group | Individualized Exercise
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individualized Exercise (N=15)
Knee pain or swelling after completing prescribed exercise that last >1 week (Musculoskeletal and connective tissue disorders) | 1 (3) — one participant reported knee pain or swelling after completing prescribed exercise that lasted more than 3 week on three separate occasions
Recurrent patellar dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) — One participant who was lost to follow-up was later found to have experienced a recurrent patellar dislocation after she finished the study intervention

LIMITATIONS AND CAVEATS:
This study was conducted at one centre and the sample size was small. Therefore, further larger-scale feasibility testing is required to determine if a full-scale randomised controlled trial comparing physiotherapy treatments for patients after acute patellar dislocation is viable

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT03798483/Prot_SAP_000.pdf